CLINICAL TRIAL: NCT06107231
Title: WHNRC (Western Human Nutrition Research Center) Honey Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: National Honey Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FL118
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Postprandial Glycemia; Metabolic Stress; Cognitive Change; Satisfaction, Personal
Keywords: Satiety; Cognition; Cortisol; Glucose; Honey; Nuts; Saliva; Stool; Almonds; Sucrose
MeSH Terms: conditions — Personal Satisfaction | interventions — Honey; Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Honey alone and honey with almonds, then sucrose alone and sucrose with almonds (Experimental): Participants will be provided honey alone once each day for 3 days, then honey plus almonds for an additional 3 days while wearing a continuous glucose monitor. After a 14 day wash-out, participants will be provided sucrose alone once each day for 3 days, then sucrose plus almonds for an additional 3 days while wearing a continuous glucose monitor.
  Interventions: Other: Honey; Other: Sucrose; Other: Honey plus almonds; Other: Sucrose plus almonds
- Sucrose alone and sucrose with almonds, then honey alone and honey with almonds (Experimental): Participants will be provided sucrose alone once each day for 3 days, then sucrose plus almonds for an additional 3 days while wearing a continuous glucose monitor. After a 14 day wash-out, participants will be provided honey alone once each day for 3 days, then honey plus almonds for an additional 3 days while wearing a continuous glucose monitor.
  Interventions: Other: Honey; Other: Sucrose; Other: Honey plus almonds; Other: Sucrose plus almonds

INTERVENTIONS:
Other: Honey — Honey representing 7% of total energy (kilocalorie) needs (40-70 grams)
Other: Sucrose — Sucrose representing 7% of total energy (kilocalorie) needs (40-70 grams)
Other: Honey plus almonds — Honey representing 7% of total energy (kilocalorie) needs (40-70 grams) plus 1 ounce almonds (28 grams)
Other: Sucrose plus almonds — Sucrose representing 7% of total energy (kilocalorie) needs (40-70 grams) plus 1 ounce almonds (28 grams)

SUMMARY:
The purpose of this research is to compare two snacks, one with honey and nuts and the other with sugar and nuts, on glucose levels before and after eating these snacks.

The investigators hypothesize that honey and nuts will have an additive effect on the reduction of postprandial glucose response. The investigators further hypothesize that consumption of honey paired with nuts will retain the benefit of sugar consumption in satiety and reduction of metabolic stress.

DETAILED DESCRIPTION:
Consuming sugar creates a feeling of satiation, and may buffer metabolic stress. However, prolonged postprandial hyperglycemia has been identified as a potential risk factor in type 2 diabetes and cardiovascular disease. Nuts, which are recommended to be consumed as part of a Mediterranean diet, up to 2 servings per day, have been shown to dramatically reduce postprandial glucose response to carbohydrates. Additionally, honey, which is typically used as an added sugar within a Mediterranean diet pattern, has a lower glycemic index than table sugar and may result in a reduced postprandial glucose response relative to other nutritive sweeteners. However, it is not yet known whether honey can work additively with nuts to further reduce postprandial glucose response over the reduction caused by nuts alone.

Honey has been shown to produce equivalent or greater satiety to regular table sugar and there is some indication that honey can improve immediate/working memory. Therefore, combined consumption of honey and nuts may offer a way to maximize the benefits of carbohydrate consumption on satiety and metabolic stress reduction while minimizing its negative effects on metabolism. However, it is not yet known whether sugars contained in the more complex food matrix of honey, consumed together with a food like nuts can impact satiety and metabolic stress in the way that has been observed for sugar.

ELIGIBILITY:
Inclusion Criteria:

* Women must be pre-menopausal
* Willing to consume snacks that contain honey, table sugar, and tree nuts

Exclusion Criteria:

* Body Mass Index (BMI) <18.5 or >40
* Allergies to tree nuts
* Current medical diagnoses of chronic diseases including cardiovascular or pulmonary diseases, renal diseases, cancer, type 1 or type 2 diabetes, thyroid disease requiring medication, inflammatory or irritable bowel diseases, or those with recent major surgeries
* No individuals who fall in to the vulnerable categories of adults including those unable to consent, pregnant women, children, or prisoners will be eligible for this study
* Routinely taking medications known to affect glucose response.
* Caffeine and alcohol use will not be excluded, but should be carefully reported by each subject.

Regarding female candidates:

* Post-menopausal
* Women who have been pregnant or nursing within the last 6 months or plan to become pregnant during the trial will be ineligible

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in postprandial glucose response | Measured continuously over days 0-8 and 23-31
  Interstitial glucose response measured by a continuous glucose monitor

SECONDARY OUTCOMES:
Change in Self-reported hunger | Fasting and 30, 60, and 90 min after consumption of standard breakfast on days 4, 8, 27, and 31
  Responses regarding hunger will be collected using a visual analog scale on a tablet with a 0-100 scale depicting the extremes (0= not at all to 100= extremely)
Change in Self-reported fullness | Fasting and 30, 60, and 90 min after consumption of standard breakfast on days 4, 8, 27, and 31
  Responses regarding fullness will be collected using a visual analog scale on a tablet with a 0-100 scale depicting the extremes (0= not at all to 100= extremely)
Change in Self-reported desire to eat | Fasting and 30, 60, and 90 min after consumption of standard breakfast on days 4, 8, 27, and 31
  Responses regarding desire to eat will be collected using a visual analog scale on a tablet with a 0-100 scale depicting the extremes (0= not at all to 100= extremely)
Change in Self-reported satisfaction with snack | Fasting and 30, 60, and 90 min after consumption of standard breakfast on days 4, 8, 27, and 31
  Responses regarding satisfaction with snack will be collected using a visual analog scale on a tablet with a 0-100 scale depicting the extremes (0= not at all to 100= extremely)
Change in Self-reported prospective consumption | Fasting and 30, 60, and 90 min after consumption of standard breakfast on days 4, 8, 27, and 31
  Responses regarding prospective consumption will be collected using a visual analog scale on a tablet with a 0-100 scale depicting the extremes (0= not at all to 100= extremely)
Change in Self-reported nausea | Fasting and 30, 60, and 90 min after consumption of standard breakfast on days 4, 8, 27, and 31
  Responses regarding nausea will be collected using a visual analog scale on a tablet with a 0-100 scale depicting the extremes (0= not at all to 100= extremely)
Change in Cognitive testing for Spatial Working Memory | Days 4, 8, 27, and 31
  Cambridge Neuropsychological Test Automated battery (CANTAB) software will be used to assess Spatial Working Memory (SWM)
Change in Cognitive testing for Paired Associates Learning | Days 4, 8, 27, and 31
  CANTAB software will be used to assess Paired Associates Learning (PAL)
Change in Cognitive testing for Rapid Visual Processing | Days 4, 8, 27, and 31
  CANTAB software will be used to assess Rapid Visual Processing (RVP)
Change in Salivary cortisol | Day 0 and 23 fasting only. Days 4, 8, 27, and 31 at fasting, 30, 60 and 90 min after consumption of snack provided in standard breakfast
  Metabolic stress will be analyzed by measuring cortisol in saliva samples
Assessment of Fasted Salivary Estradiol | Days 0, 4, 8, 23, 27,and 31 at fasting only
  Passive drool will be assayed for estradiol as they impact metabolic stress throughout study days
Assessment of Fasted Salivary Progesterone | Days 0, 4, 8, 23, 27,and 31 at fasting only
  Passive drool will be assayed for progesterone as they impact metabolic stress throughout study days
Change in Stool marker of inflammation | Stool collected on study days 0, 4, 8, 23, 27, and 31
  Fecal calprotectin measured in stool samples
Change in Stool bacterial metagenomics | Stool collected on study days 0, 4, 8, 23, 27, and 31
  Honey responsive genes identified by metagenomics
Change in Dietary Intake | Days 1-3, 5-7, 24-26, and 28-30
  Food records collected using Automated Multi-pass Method (AMPM) on the platform ASA24

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kable, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center; Nancy Keim, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center; Kevin Laugero, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Background] Anderson GH, Woodend D. Consumption of sugars and the regulation of short-term satiety and food intake. Am J Clin Nutr. 2003 Oct;78(4):843S-849S. doi: 10.1093/ajcn/78.4.843S. PMID 14522748
- [Background] Tryon MS, Stanhope KL, Epel ES, Mason AE, Brown R, Medici V, Havel PJ, Laugero KD. Excessive Sugar Consumption May Be a Difficult Habit to Break: A View From the Brain and Body. J Clin Endocrinol Metab. 2015 Jun;100(6):2239-47. doi: 10.1210/jc.2014-4353. Epub 2015 Apr 16. PMID 25879513
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Gallwitz B. Implications of postprandial glucose and weight control in people with type 2 diabetes: understanding and implementing the International Diabetes Federation guidelines. Diabetes Care. 2009 Nov;32 Suppl 2(Suppl 2):S322-5. doi: 10.2337/dc09-S331. No abstract available. PMID 19875573
- [Background] Bach-Faig A, Berry EM, Lairon D, Reguant J, Trichopoulou A, Dernini S, Medina FX, Battino M, Belahsen R, Miranda G, Serra-Majem L; Mediterranean Diet Foundation Expert Group. Mediterranean diet pyramid today. Science and cultural updates. Public Health Nutr. 2011 Dec;14(12A):2274-84. doi: 10.1017/S1368980011002515. PMID 22166184
- [Background] Josse AR, Kendall CW, Augustin LS, Ellis PR, Jenkins DJ. Almonds and postprandial glycemia--a dose-response study. Metabolism. 2007 Mar;56(3):400-4. doi: 10.1016/j.metabol.2006.10.024. PMID 17292730
- [Background] Larson-Meyer DE, Willis KS, Willis LM, Austin KJ, Hart AM, Breton AB, Alexander BM. Effect of honey versus sucrose on appetite, appetite-regulating hormones, and postmeal thermogenesis. J Am Coll Nutr. 2010 Oct;29(5):482-93. doi: 10.1080/07315724.2010.10719885. PMID 21504975
- [Background] Gourdomichali T, Papakonstantinou E. Short-term effects of six Greek honey varieties on glycemic response: a randomized clinical trial in healthy subjects. Eur J Clin Nutr. 2018 Dec;72(12):1709-1716. doi: 10.1038/s41430-018-0160-8. Epub 2018 Apr 24. PMID 29686412
- [Background] Othman Z, Shafin N, Zakaria R, Hussain NH, Mohammad WM. Improvement in immediate memory after 16 weeks of tualang honey (Agro Mas) supplement in healthy postmenopausal women. Menopause. 2011 Nov;18(11):1219-24. doi: 10.1097/gme.0b013e31821e2044. PMID 21926932
- [Background] Gonzalez-Rodriguez M, Pazos-Couselo M, Garcia-Lopez JM, Rodriguez-Segade S, Rodriguez-Garcia J, Tunez-Bastida C, Gude F. Postprandial glycemic response in a non-diabetic adult population: the effect of nutrients is different between men and women. Nutr Metab (Lond). 2019 Jul 17;16:46. doi: 10.1186/s12986-019-0368-1. eCollection 2019. PMID 31346341
- [Background] Carroll JF, Kaiser KA, Franks SF, Deere C, Caffrey JL. Influence of BMI and gender on postprandial hormone responses. Obesity (Silver Spring). 2007 Dec;15(12):2974-83. doi: 10.1038/oby.2007.355. PMID 18198306
- See also: CDC National Diabetes Statistics Report, 2020, Estimates of Diabetes and Its Burden in the United States — https://www.cdc.gov/diabetes/php/data-research/?CDC_AAref_Val=https://www.cdc.gov/diabetes/pdfs/data/statistics/national-diabetes-statistics-report.pdf

DOCUMENTS (1):
  • Informed Consent Form (2025-05-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT06107231/ICF_000.pdf